CLINICAL TRIAL: NCT03369041
Title: Study of the Practice of Debiri in France: Indications, Associations to Systemic Treatments, Efficiency, Tolerance - Prospective Practice Survey
Brief Title: Study of the Practice of Debiri in France
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Other Study IDs: DEBIRI Cohort
Record Dates: First submitted 2017-07-13; First posted 2017-12-11 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Adenocarcinoma; Hepatic Metastases
Keywords: chemoembolization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Irinotecan-Eluting Beads
  Other Names: DEBIRI

SUMMARY:
In order to extract the profiles of patients receiving DEBIRI treatment at best, the investigators proposed the establishment of a national prospective cohort to collect information on the greatest number of patients treated with DEBIRI. This cohort will allow a better understanding of the effectiveness, tolerance, feasibility and differences of practices at national level for this approach. These data will assist in the development of clinical trials in situations that appear to be most promising in clinical practice.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer in men and the second in women (1.23 million cases in 2008, 608700 deaths) 40 to 50% of patients developed hepatic, synchronous or metachronous metastases. In 10 to 15% of cases, these metastases are operable initially, and a perioperative chemotherapy of the FOLFOX type is then most performed. In about 20% of patients discharged metastases resectable after induction chemotherapy. When hepatic invasion makes a complete resection impossible, a palliative treatment is initiated, mainly based on chemotherapy with or without biotherapies (anti-VEGF or anti-EGFR).

In recent years, intra-hepatic arterial treatments have been developed, with the aim of improving the prognosis of inoperable patients. The particular vascular anatomy of the liver makes it possible to perform local work via its main artery or its branches. The hepatic artery provides 25% of the blood flow and 50% of the oxygenation of the liver, the portal vein ensures 75% of the blood flow and also 50% of the oxygenation. Primary or secondary tumors are mainly focused on the artery and the rest of the parenchyma mainly through the portal vein, treatment of tumors using the arterial route also allows to administer under satisfactory safety conditions the therapeutic agent of Many More selective within the tumor, saves healthy hepatic tissue.

Several approaches to intra-arterial treatments have been developed to date, such as hepatic intra-arterial chemotherapy, radioembolization, or micro-bead embolization (DC-Beads®). In the latter case, they are DEB Drug Eluting Beads at irinotecan, in the context of a treatment called DEBIRI. Thanks to their diameter of 75 to 300 μm, they allow embolization of the tumor's arterioles, with a dual objective: to create tumor ischemia and increase the intra-tumor concentration in chemotherapy. The advantage of this approach is simplicity. Contrary to the two previous techniques (radio and chemo-embolization), it does not require the placement of an intra-arterial catheter, nor the administration of a radioactive agent imposing heavy use constraints. It could make this intra-arterial technique accessible in many centers and thus benefit a greater number of patients.

Data on the use of this strategy remain limited, and concern patients already treated by several lines of chemotherapy. The response rates in these heavily pretreated patients are encouraging.

Several questions arise: firstly, what is the place of this treatment used so far in patients treated with the treatises (2 tests currently published). In practice, few patients have limited liver disease after 2 or 3 lines of chemotherapy, which reserves this approach for a small minority of patients. It should be tried to develop this technique earlier in the cost of patients, in order to propose, for example, as a consolidation treatment in patients who are not resectable or to try to have a down-sizing in potentially resectable patients. Response rate of 65% in pretreated patients.

Other questions remain unanswered about this therapeutic approach: should systemic treatment with 5FU be used to reduce the risk of extrahepatic progression? Is it possible, and can the investigators associate, systemic chemotherapy such as oxaliplatin to intensify the response? And finally, what is the place of biotherapies in this strategy? None of the questions have been discussed with DEBIRI to date.

In order to extract the profiles of patients receiving DEBIRI treatment at best, the investigators propose the establishment of a national prospective cohort to collect information on the greatest number of patients treated with DEBIRI. This cohort has allowed a better understanding of the effectiveness, tolerance, feasibility and differences of practices at national level for this approach. These data will assist in the development of clinical trials in situations that appear to be most promising in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Histologically proven colorectal adenocarcinoma
* Synchronous or metachronous hepatic metastases
* No significant extrahepatic disease
* Indication of treatment by DEBIRI retained
* Patient who received the information note

Exclusion Criteria:

* Patients who started treatment with DEBIRI before 2015
* Patients who for psychological, social, family or geographic reasons could not be monitored regularly.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven colorectal adenocarcinoma and synchronous or metachronous hepatic metastases with indication of treatment by DEBIRI retained after 2015.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) and/or hepatic progression free survival | 3 years after inclusion

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years after inclusion
Best response rate | 6 months after the end of treatment

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Centre Hospitalier de Blois, Blois
  - Avicenne, Bobigny
  - CHU Estaing, Clermont-Ferrand
  - Clinique des Cèdres, Cornebarrieu
  - Centre Hospitalier Intercommunal St. Aubin les Elbeuf, Elbeuf
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - CHU de Grenoble, Grenoble
  - Centre Léon Berard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Le Raincy Montfermeil, Montfermeil
  - Centre Antoine Lacassagne, Nice
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - Hôpital de la Miletrie, Poitiers
  - CH, Reims
  - HIA Begin, Saint-Mandé

IPD SHARING:
Plan to Share IPD: Undecided